CLINICAL TRIAL: NCT01399255
Title: Comparative Bioequivalence Study of Wockhardt's Insulin Analogue Lispro (Listro™) With Humalog® in Healthy Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was not initiated
Sponsor: Wockhardt (Industry)
Responsible Party: Dr.R Jha ,Senior Vice-president - Clinical Research, Wockhardt Limited
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: Listro/PK-PD/FDA/2011
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Bioequivalence in Healthy Subjects
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Listro™ Arm (Experimental): Insulin Lispro (Listro™); 100 U/mL, DispoPen 3.0 mL.
  Interventions: Biological: Insulin lispro
- Humalog® Arm (Active Comparator): Insulin Lispro (Humalog®; 100 U/mL), Humalog® Kwik Pen™ 3.0 mL.
  Interventions: Biological: Insulin lispro

INTERVENTIONS:
Biological: Insulin lispro — Dosage form- Subcutaneous Injection
  Other Names: Listro™ and Humalog®

SUMMARY:
The aim of this study is to assess the bioequivalence of two rapid-acting insulin Lispro formulations: Humalog® and Listro™ in healthy subjects based on the pharmacokinetic parameter (PK) and the pharmacodynamic parameter (PD).

DETAILED DESCRIPTION:
The purpose of this study is to assess the bioequivalence of two rapid-acting insulin Lispro formulations: Humalog® and Listro™ in healthy subjects, based on the pharmacokinetic parameter (PK) AUC (INS-LIS 0-8h) and the pharmacodynamic parameter (PD) AUC (GIR 0-8h) and also assess the safety and local tolerability of the two insulin preparations.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects.
2. Age ≥18 and ≤50 years.
3. Considered generally healthy upon completion of medical history, physical examination and biochemical investigations as judged by the Investigator.
4. Body Mass Index (BMI) between 18.0 and 27.0 kg/m2, inclusive.
5. Non-smoker, defined as no nicotine consumption for at least one year.
6. Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject)

Exclusion Criteria:

1. Previous participation in this trial or other clinical trials within the last 30 days.
2. Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures (e.g. intrauterine device (IUD) that has been in place for at least 3 months, or sterilization, or the oral contraceptive pill, which should have been taken without difficulty for at least 3 months, an approved hormonal implant or double barrier method) including male condoms used plus spermicide, diaphragm with spermicide plus male condom cap with spermicide plus male condom are acceptable options).
3. Clinically significant abnormal hematology or biochemistry screening tests, as judged by the Investigator. In particular, subjects with an elevated fasting blood glucose, elevated liver enzymes (AST or ALT >2 times the upper limit of normal) or impaired renal function (elevated serum creatinine values above the upper limit will not be allowed to enter the trial. Subjects with abnormal TSH may be required to have additional testing of thyroid hormones for further clarification. Subjects with abnormal TSH judged by the Investigator as clinically significant will be excluded from the study.
4. Any serious systemic infectious disease during the four weeks prior to the first dose of test drug, as judged by the Investigator.
5. History of any illness that, in the opinion of the Investigator, might confound the results of the trial or pose risk in administering the trial drug to the subject. In particular, subjects with significant cardiovascular disease, anemia (hemoglobin below the lower limit of normal) or hemoglobinopathy will not be allowed to enter the trial.
6. Cardiac problems defined as decompensated heart failure (New York Heart Association (NYHA) class III and IV) at any time and/or angina pectoris within the last 12 months and/or acute myocardial infarction at any time.
7. Clinically significant abnormal ECG at screening, as judged by the Investigator.
8. History of alcohol or drug abuse in the past five years.
9. Any positive screen for drugs of abuse.
10. Hepatitis B or C or HIV positive.
11. Use of prescription drugs within 3 weeks preceding the first dosing of insulin, except for oral contraceptives/hormonal implants.
12. Use of non-prescription drugs, except routine vitamins or herbal products, within 3 weeks prior to the first dose of the test drug.
13. Occasional use of acetaminophen is permitted. Acetaminophen is not allowed on the dosing day until 4 hours postdosing.
14. Use of systemic corticosteroids, monoamine oxidase (MAO) inhibitors, prostaglandin blockers, systemic non-selective beta-blockers, growth hormones
15. Thyroid hormones are not allowed unless stable during the past 3 months.
16. Any use of non-steroid anti-inflammatory drugs (NSAIDs) except for low-dose Aspirin is not allowed within 7 days prior to dosing and on the dosing day.
17. Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation.
18. Blood donation of more than 500 ml within the last 12 weeks.
19. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
20. Known or suspected allergy to trial product or related products.
21. History of deep leg vein thrombosis or a frequent appearance of deep leg vein thrombosis in 1st degree relatives (parents, siblings or children) as judged by the Investigator.
22. Any disease or condition that, in the opinion of the Investigator, would represent an unacceptable risk for the subject's safety.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence based on Pharmacokinetic parameter AUC (INS-LIS 0-8h) | 8 hrs post dose
  Glucose clamp will be terminated 10 hours post dose and the primary pharmacokinetic bioequivalance will be calculated based on the Area under the curve (AUC) between 0 - 8 hours postdose of the study medication.
Bioequivalence based on Pharmacodynamic parameter: AUC (GIR 0-8h) | 8 hrs post dose
  Glucose clamp will be terminated 10 hours post dose and the primary pharmacodymanic bioequivalance will be calculated based on the Area under the curve (AUC) for the glucose infusion rate (GIR) between 0 - 8 hours postdose of the study medication

SECONDARY OUTCOMES:
Pharmacokinetic parameters:Maximum concentration (Cmax) | over 10 hrs post dose
Pharmacodynamic parameters: Area under curve glucose infusion rate from 0-10hrs | over 10 hrs post dose
  AUC (GIR 0-4h), AUC (GIR 4-8h), AUC (GIR 4-10h), AUC (GIR 0-10h)
Safety endpoints | over 10 hrs post dose
  Number of AE's, SAE's, Hypoglycemic events and local tolerability
Pharmacokinetic parameter: Area under curve from 0-10hrs | over 10 hours postdose
  AUC (INS-LIS 0-4 h), AUC (INS-LIS 4-8 h), AUC (INS-LIS 4-10h), AUC (INS-LIS 0-10 h)
Pharmacokinetic Parameters: tmax and t1/2 | Over 10 hours postdose
Pharmacodynamic parameter: GIR max and tGIR max | over 10 hrs postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Profil Institute for Clinical Research, Inc., Chula Vista, California, United States